CLINICAL TRIAL: NCT00515112
Title: A Randomized, Double Blind, Placebo-Controlled Phase II Study of Testosterone Replacement in Men With Non-Metastatic Castrate Resistant Prostate Cancer
Brief Title: Testosterone Replacement in Men With Non-Metastatic Castrate Resistant Prostate Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: This study has been terminated due to poor accrual
Sponsor: University of Chicago (Other)
Collaborators: Solvay Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 15393B
Record Dates: First submitted 2007-08-09; First posted 2007-08-13 (Estimated); Results first posted 2014-06-11 (Estimated); Last update posted 2014-06-11 (Estimated); Status verified 2014-05

CONDITIONS: Prostate Cancer
Keywords: prostate; cancer; testosterone replacement; AndroGel; prostatic cancer; prostatic neoplasms
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasms | interventions — Testosterone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Experimental): Twenty subjects will receive testosterone gel
  Interventions: Drug: AndroGel
- B (Placebo Comparator): Twenty subjects will receive the placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: AndroGel — Androgel 1%, 10g daily
  Arms: A
Drug: placebo — placebo
  Arms: B

SUMMARY:
The purpose of this study is to determine whether prostate cancer growth can be slowed in patients who receive Androgel® 1% at 10 gram dose.

DETAILED DESCRIPTION:
The primary objective of the study is to determine the effect of testosterone replacement on time to disease progression and time to clinical cancer progression.

The secondary objectives are to describe the effect of testosterone replacement on patient-reported quality of life (FACT-P, FACT-fatigue and specific measures from the Expanded Prostate Cancer Index (EPIC): Sexual and Hormonal Assessments), and hand-grip strength; to describe changes in total testosterone, free testosterone, and PSA levels; to explore AR levels in circulating tumor cells as a marker of treatment benefit.

ELIGIBILITY:
Inclusion Criteria:

* Prostate cancer
* Patient must have received primary definitive local therapy to the prostate (surgery and/or radiotherapy)
* Patient was surgically or pharmacologically castrated at least 6 months prior to starting the study
* Patient must have had a previous trial of anti-androgen therapy
* Patient must have a rising PSA
* No evidence of distant metastatic disease
* ECOG performance status < 2
* Age >18 years
* Patients must have normal hepatic function

Exclusion Criteria:

* Patients with a history of any previous cytotoxic therapy or radionuclide therapy (such as rhenium, strontium, or samarium)
* Patients may not be receiving any other investigational agents
* Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, uncontrolled cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Patients receiving renal dialysis
* Patients with significant pulmonary disease who have received chronic or pulse steroid therapy within the last 3 months prior to randomization will be excluded
* Patients who have known hypersensitivity to any of the AndroGel ingredients, including testosterone that is chemically synthesized from soy

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2007-07; Primary Completion 2010-11 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Walter Stadler, MD, Principal Investigator — University of Chicago
Locations (11):
- United States (11):
  - University of Southern California, Los Angeles, California
  - University of Colorado, Aurora, Colorado
  - Northwestern University, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - NorthShore University Helath System, Evnaston, Illinois
  - Ingalls Memorial Hospital, Harvey, Illinois
  - Illinois Cancer Care, Peoria, Illinois
  - University of Maryland, Baltimore, Maryland
  - University of Rochester, Rochester, Maryland
  - Baylor College of Medicine, Houston, Texas
  - Medical College of Wisconsin, Milwaukee, Wisconsin

REFERENCES:
- [Derived] Geynisman DM, Szmulewitz RZ, Stadler WM. A trial postmortem: challenges in conducting a randomized, double-blind, phase 2 study in men with castration-resistant prostate cancer. Eur Urol. 2012 Nov;62(5):864-6. doi: 10.1016/j.eururo.2012.08.030. Epub 2012 Aug 25. No abstract available. PMID 22939385

RESULTS

PARTICIPANT FLOW:
Groups:
- Androgel: Three subjects received testosterone gel
  AndroGel: Androgel 1%, 10g daily
- Placebo: Three subjects received the placebo
  Placebo: placebo
Period: Overall Study
Arm/Group | Androgel | Placebo
Started | 3 | 3
Completed | 0 | 0
Not Completed | 3 | 3
Not completed — Death | 0 | 1
Not completed — The study was terminated | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Androgel | Placebo | Total
Number analyzed (Participants) | 3 | 3 | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.4 (4.6) | 63.5 (8.6) | 66.4 (7.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 3 | 3 | 6

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival
Description: Time to progression is measured from the date of randomization until the onset of the earliest of one of the following events: in the absence of a 50% decline in prostate-specific antigen (PSA), a PSA increase to 3 times the nadir PSA or an absolute PSA value of 50 ng/ml, whichever comes first; if at least a 50% decline in PSA is achieved from PSA peak value, a PSA increase of 50% above the nadir provided the increase is at least 5 ng/ml or back to baseline; one or more new skeletal lesions as shown on any bone scan or minimum of 1.5 cm in longest diameter on any computed tomography or magnetic resonance imaging scan; tumor flair; the occurrence of a clinical event, including death, determined by the investigator to represent disease progression.
Time Frame: Up to 5 years
Population: This study has been terminated due to poor accrual.
Arm/Group | Androgel | Placebo
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: To Explore the Value of Androgen Receptor (AR) Expression in Circulating Tumor Cells.
Description: The AR is defined as 4 categories by the observed data: no detectable cells, low AR expression, normal AR expression, and high AR expression.
Time Frame: every 8 weeks
Arm/Group | Androgel | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Androgel | Placebo
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Androgel (N=3) | Placebo (N=3)
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Alkaline phosphatase increased (Investigations) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Blood bicarbonate decreased (Investigations) | 1 | 0
Coarse hair (Skin and subcutaneous tissue disorders) | 1 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 0
Dark stools (Gastrointestinal disorders) | 0 | 1
Erectile dysfunction (Reproductive system and breast disorders) | 0 | 1
Fatigue (General disorders) | 1 | 1
Hemoglobin (Investigations) | 2 | 1
Hemoglobin decreased (Investigations) | 1 | 1
Hemorrhage urinary tract (Renal and urinary disorders) | 0 | 1
Hyperglycemia (Investigations) | 0 | 1
Hyperkalemia (Investigations) | 0 | 1
Hypokalemia (Metabolism and nutrition disorders) | 0 | 2
Hypophosphatemia (Investigations) | 0 | 1
Insomnia (Psychiatric disorders) | 1 | 0
Joint pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Libido decreased (Psychiatric disorders) | 1 | 0
Lymphopenia (Investigations) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Pain- other: shoulder and back pain (General disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
Urinary frequency (Renal and urinary disorders) | 1 | 1
Urogenital disorder (Renal and urinary disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No